CLINICAL TRIAL: NCT02475564
Title: The Use of Resveratrol for Pain in Endometriosis - A Clinical Trial
Brief Title: Resveratrol for Pain Due to Endometriosis
Acronym: ResvEndo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 140626
Record Dates: First submitted 2015-06-11; First posted 2015-06-18 (Estimated); Results first posted 2016-08-05 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-08

CONDITIONS: Endometriosis
Keywords: resveratrol
MeSH Terms: conditions — Endometriosis | interventions — Starch; Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Patients will take once a day a monophasic pill (ethinylestradiol + levonorgestrel) continuously for 42 days with 1 pill of placebo (starch)
  Interventions: Drug: Placebo
- resveratrol (Experimental): Patients will take once a day a monophasic pill (ethinylestradiol + levonorgestrel) continuously for 42 days with 40mg of resveratrol
  Interventions: Drug: Resveratrol

INTERVENTIONS:
Drug: Placebo — 40mg of starch
  Other Names: Starch
  Arms: placebo
Drug: Resveratrol — 40mg of resveratrol (powder)
  Arms: resveratrol

SUMMARY:
This study aims to verify whether the use of 40 mg of resveratrol per day associated with monophasic contraceptive pill (levonorgestrel 0.15mg/ethinyl estradiol 0.03mg) reduces pelvic pain at the end of 2 months of treatment, compared to the use of the pill with placebo.

DETAILED DESCRIPTION:
Endometriosis is a disease that affects 176 million women around the world, and it is present in about 60% of adolescent women with chronic pelvic pain and dysmenorrhea. Some researchers have investigated the antiproliferative effect of resveratrol in endometriosis using animal models and humans. The reduction in the size and activity of the endometriotic implants has been observed with the use of resveratrol. The reduction of pain in patients with endometriosis is an important aspect of the quality of life. The use of a medication with few side effects and the lack of clinical quality trials justify this study, which aims to verify whether the use of 40 mg of resveratrol per day associated with monophasic contraceptive pill reduces pelvic pain at the end of 2 months of treatment, compared to the use of the pill with placebo. This study will be randomized, prospective, double blind with two arms of 22 patients; the CONSORT parameters will be followed. The degree of pain by visual analog scale, prolactin levels (ng / mL) and the carcinoembryonic antigen levels (CA125) (IU / L) will be measured at the begging and at the end of trial. These parameters will be the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Endometriosis diagnosed by laparoscopy

Exclusion Criteria:

* Known allergy to resveratrol
* Use of gonadotropin or danazol in the last month

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Savaris, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- HCPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Johnson NP, Hummelshoj L; World Endometriosis Society Montpellier Consortium. Consensus on current management of endometriosis. Hum Reprod. 2013 Jun;28(6):1552-68. doi: 10.1093/humrep/det050. Epub 2013 Mar 25. PMID 23528916
- [Result] Amaya SC, Savaris RF, Filipovic CJ, Wise JD, Hestermann E, Young SL, Lessey BA. Resveratrol and endometrium: a closer look at an active ingredient of red wine using in vivo and in vitro models. Reprod Sci. 2014 Nov;21(11):1362-9. doi: 10.1177/1933719114525271. Epub 2014 Mar 6. PMID 24604232
- [Result] Maia H Jr, Haddad C, Pinheiro N, Casoy J. Advantages of the association of resveratrol with oral contraceptives for management of endometriosis-related pain. Int J Womens Health. 2012;4:543-9. doi: 10.2147/IJWH.S36825. Epub 2012 Oct 10. PMID 23091400

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 18th and November 6th, 2015, 234 women with diagnosis of endometriosis were screened for the study at outpatient clinic of Hospital de Clínicas de Porto Alegre, Porto Alegre, RS, Brazil
Period: Overall Study
Arm/Group | Placebo | Resveratrol
Started | 22 | 22
Completed | 18 | 21
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Intense Menstrual bleeding | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resveratrol | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (7.1) | 32.4 (7) | 33.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  white | 16 | 15 | 31
  black | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  Brazil | 22 | 22 | 44
Baseline pain levels (Visual Analog Scale - VAS) day 1 [Mean (Standard Deviation); unit: units on a scale] — A 10 cm slide ruler, marked at regular intervals in millimeters, was used for measuring pain intensity on a Visual Analog Scale. The scale had scores ranging continuously from 0 (no pain) to 10 (worst imaginable pain).
  units on a scale | 5.4 (2.6) | 5.7 (2) | 5.6 (2.3)
CA-125 [Median (Full Range); unit: UI/mL] | 14.1 [3.3 to 49.5] | 18.7 [5.7 to 123.6] | 17.04 [3.3 to 123.6]
Prolactin [Mean (Standard Deviation); unit: ng/mL] | 12.65 (5.9) | 14.27 (6.6) | 13.13 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores Measured by VAS (Visual Analog Scale) at Day 42.
Description: Pain will be measured by VAS (visual analog scale) as baseline and at the end of the study, considering the last 7 days. VAS was used to measuring pain intensity, ranging continuously from 0 (no pain) to 10 (worst imaginable pain). The main outcome compared median pain levels between both arms on day 42.
Time Frame: 42 days
Population: Intention to treat analysis, patients who were lost on follow-up had their last registry on pain values or plasma levels measurements repeated in the following consultations.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 22 | 22
units on a scale | 3.2 [0 to 8] | 3.9 [0 to 8.9]
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; A sample size of at least 21 patients per arm would be necessary to have a 90% chance of detecting, as significant at the 1% level, a difference of 3 points in a scale of 10 points, between both groups as the primary outcome, after 42 days of treatment; Test type: Superiority or Other; p = 0.7, Mann-Whitney test

2. Secondary Outcome: Serum CA125 Levels at 42 Days
Description: Serum levels of CA125 will be measured after 42 days of treatment in UI/mL. Median levels of CA125 were compared between both groups on day 42, and to baseline values (day 1).
Time Frame: 42 days
Population: One of subjects from the placebo group decided to leave the study after randomization, thus the n = 21 in the CA125 levels.
Measure: Median (Full Range); unit: UI/mL
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 22 | 21
UI/mL | 11.7 [4.9 to 29.9] | 13.7 [5 to 61]
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.1, Mann-Whitney test

3. Secondary Outcome: Serum Prolactin Levels at 42 Days
Description: Serum levels of prolactin will be measured after 42 days of treatment. Median levels of prolactin were compared between both groups on day 42.
Time Frame: 42 days
Population: one of the subjects in the placebo group decided to leave the study after randomization, thus n = 21
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Resveratrol | Placebo
Number analyzed (Participants) | 22 | 21
ng/mL | 12 [4.3 to 32.1] | 11.1 [4.2 to 31.6]
Statistical Analysis 1: Comparison: Resveratrol vs Placebo; Test type: Superiority or Other; p = 0.8, Mann-Whitney test

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Placebo | Resveratrol
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 10/22 | 13/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Resveratrol (N=22)
headache (Nervous system disorders) | 7 (7) | 6 (6) — 6 cases of mild headache
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Reduced libido (Reproductive system and breast disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hot flushes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Increased uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
candidiasis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
dispareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
There were only 42 days of treatment observed, a longer follow-up, for instance 6 months, may impact the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No